CLINICAL TRIAL: NCT05609903
Title: Atezolizumab in Combination With Nab-paclitaxel for Patients With Previously Untreated Metastatic Triple-negative Breast Cancer in a Real World Experience
Brief Title: Atezolizumab With Nab-paclitaxel for Patients With Triple-negative Stage IV Breast Cancer
Acronym: Anastase
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID4060
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer Metastatic
Keywords: Atezolizumab; Nab-Paclitaxel, Metastatic Breast Cancer;
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Atezolizumab in combination with nab-paclitaxel — Treatment of patients with stage IV triple negative breast cancer with Atezolizumab in combination with nab-paclitaxel

SUMMARY:
The study will evaluate the therapeutic efficacy of the association of Atezolizumab plus nabPaclitaxel in a real life context, in order to document any differences both in terms of activity and safety with respect to the knowledge of the association reported in the literature

DETAILED DESCRIPTION:
On 8thMarch 8 2019, the Food and Drug Administration (FDA) granted accelerated approval to Atezolizumab in combination with nab-paclitaxel for adult patients with unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) whose tumors express PD-L1 (PD-L1 stained tumor-infiltrating immune cells [IC] of any intensity covering ≥ 1% of the tumor area). FDA also approved the Ventana PD-L1 (SP142) Assay as a companion diagnostic device for selecting TNBC patients for atezolizumab. Approval was based on the clinical trial IMpassion130 results.

In EU, the Committee for Medicinal Products for Human Use (CHMP) issued positive opinion on 27thJune 2019 for the use of Atezolizumab 840 mg in combination with nab-paclitaxel for the treatment of adult patients with unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) whose tumours have PD-L1 expression ≥ 1% and who have not received prior chemotherapy for metastatic disease. Hereafter, the European Commission approved Atezolizumab for the treatment of mTNBC in August 2019.

In some cases, free access to pharmaceutical treatment is allowed in Italy before AIFA authorises its marketing or, for medicines already authorised, for indications other than those for which the medicinal product has been authorised in Italy (off-label use). One route for early access to a medicinal product is Compassionate use that involves direct and free delivery of the medicine by the manufacturer.

Due to the severity of the disease and the lack of further valid therapeutic alternatives, Roche S.p.A. in accordance with AIFA opened a Compassionate Use Program (CUP) based on the European indication mentioned above on 18th November 2019. The Program closed on 28th August 2020 following the approval and reimbursement granted by AIFA to Atezolizumab in mTNBC.

To date the drug is therefore available and reimbursed by the national health system, and has become part of daily clinical practice, as also indicated by the most recent AIOM guidelines.

Randomized controlled trials (RCTs) are trials in selected patients, they have a high internal validity but low external validity, their results could not extend to real word patient with different characteristics (patients in more severe or less severe clinical conditions, protected bands), there are a few data on interactions with concomitant diseases and therapies and on actual compliances with other therapies.

Real world evidence is important as it complements data from RCTs. After the pivotal trial, it is essential to continue studying the risk-benefit profile of the combination and therefore it is necessary carry out real world experience.

In the context of Compassionate Use Program a hundred patients have been treated with Atezolizumab plus nab-paclitaxel throughout Italy and it would be scientifically interesting to collect their data retrospectively as the first source of efficacy and safety of this combination in a real population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years who have provided written informed consent
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* No prior chemotherapy, experimental or targeted systemic therapy for inoperable locally advanced or metastatic TNBC. Prior chemotherapy (including taxanes) in the neoadjuvant or adjuvant setting is allowable if treatment was completed ≥12 months prior to enter the compassionate use program
* PD-L1-positive tumour status defined as PD-L1 expression ≥1% on tumour-infiltrating immune cells as percentage per tumour area, assessed by the Ventana PD-L1 (SP142) assay based on the status of the primary tumor and/or the biopsy of metastatic disease before starting the treatment. Samples should be assessed by a qualified laboratory and different assays are not acceptable
* Patients eligible for ongoing atezolizumab clinical trials from which they may benefit are excluded
* Eligible for taxane monotherapy (i.e., absence of rapid clinical progression, life-threatening visceral metastases, or the need for rapid symptom and/or disease control)
* ECOG performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1)
* ANC ≥1500 cells/µL (without granulocyte colony-stimulating factor [G-CSF] support within 2 weeks prior to Cycle 1, Day 1);
* Lymphocyte count ≥500/µL; Platelet count ≥100,000/µL (without transfusion within 2 weeks prior to Cycle 1, Day 1);
* Hemoglobin ≥9.0 g/dL; AST, ALT, and alkaline phosphatase ≤2.5x the upper limit of normal (ULN), with the following exceptions:
* Patients with documented liver metastases: AST and ALT ≤5x ULN
* Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5x ULN
* Serum bilirubin ≤1.25x ULN (patients with known Gilbert disease who have serum bilirubin level ≤3x ULN may be enrolled)
* INR and aPTT ≤1.5x ULN (this applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose)
* Calculated creatinine clearance ≥30 mL/min
* Absence of a positive test for HIV, active hepatitis B or hepatitis C, active tuberculosis
* Absence of significant cardiovascular disease (New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to treatment start, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) <40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate)
* No known untreated, symptomatic or corticosteroid-dependent brain metastases
* Patients with any history of immune deficiencies or autoimmune disease are excluded from the treatment. Possible exceptions could be autoimmune-mediated hypothyroidism on a stable dose of thyroid replacement hormone, controlled type 1 diabetes mellitus on a stable insulin dosing regimen, eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only
* Patients must not be administered systemic immunostimulatory agents within 4 weeks or systemic immunosuppressive medications within 2 weeks prior to start the treatment
* Patients must agree not to receive live, attenuated vaccine (e.g., FluMist®) within 28 days prior to the first dose of study treatment (Cycle 1, Day 1), during treatment, or within 5 months following the last dose of atezolizumab
* No known hypersensitivity or allergy to nab-paclitaxel, to any of the excipients, to biopharmaceuticals produced in Chinese hamster ovary cells, or to any component of the atezolizumab formulation
* Pregnancy or lactation are general medical exclusion criteria from the treatment
* Women of child bearing potential must agree to either use a contraceptive method with a failure rate of ≤ 1% per year or to remain abstinent (refrain from heterosexual intercourse) during the treatment period and for at least 5 months after the last dose of atezolizumab or 1 month after the last dose of nab-paclitaxel, whichever is later. For definition of postmenopausal status see the study protocol
* Women of child bearing potential must have a negative serum pregnancy test result prior to start the treatment

Esclusion Criteria:

* Patients who have not completed 1 cycle of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged ≥ 18 with biopsy proven Triple Negative Breast Cancer locally advanced or stage IV at diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Objective responce rate | 1 year
  Rate of patients with a partial responce or stable disease
Time-to-treatment discontinuation | 1 year
  Time from tha start of therapy to the time of treatment discontinuation for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Policlinico A. Gemelli
Locations (1):
- Policlinico A. Gemelli - IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No